CLINICAL TRIAL: NCT03042351
Title: Pilot Study for the Urinary Incontinence Treatment by Using a Pelvic Floor Muscles Restorative Device (E-NNA®)
Brief Title: Pilot Study for the Urinary Incontinence Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Palacios (Other)
Collaborators: eCareYou Innovation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-ENNA-2015
Record Dates: First submitted 2016-10-04; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Pelvic Floor
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Unique arm (Other): Magic Kegel app
  Interventions: Device: Magic Kegel app

INTERVENTIONS:
Device: Magic Kegel app — Pelvic floor muscles recover exercises with a specific device and Magic Kegel App

SUMMARY:
Non invasive study to improve the urinary incontinence, through pelvic floor muscles exercises

DETAILED DESCRIPTION:
A non invasive study to improve the urinary incontinence performed in 36 women from two groups: 18 menopausal women and 18 fertile women. The participants have to do pelvic floor muscles exercises with a restorative pelvic floor device every day for two months using the Magic Kegel app download in their mobile devices

ELIGIBILITY:
Inclusion Criteria:

* Urinary incontinence diagnosis

Exclusion Criteria:

* No urinary infection
* No surgery for urinary incontinence

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Changes in values registered in Magic Kegel App | Six months

SECONDARY OUTCOMES:
Changes in ICIQ-SF questionnaire at month 2 respect to baseline | 60 days
Changes in FSFI questionnaire at month 2 respect to baseline | 60 days
Changes in Sandvick questionnaire at month 2 respect to baseline | 60 days
Changes in PISQ-12 questionnaire at month 2 respect to baseline | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Palacios, MD, Principal Investigator — Instituto Palacios
Locations (1):
- Instituto Palacios, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No